CLINICAL TRIAL: NCT05734846
Title: Biofinity Multifocal Contact Lenses Fitting Methods Comparison
Brief Title: Multifocal Contact Lenses Fitting Methods Comparison
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-22-49
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Results first posted 2024-01-10 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2023-02

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Lenses, then Test Lenses (Experimental): Participants wore the Control Lenses for 1 week, then crossed over to the Test Lenses for 1 week.
  Interventions: Device: Control Lenses (control fitting approach); Device: Test Lenses (test fitting approach)
- Test Lenses, then Control Lens (Experimental): Participants wore the Test Lenses for 1 week, then crossed over to the Control Lenses for 1 week.
  Interventions: Device: Control Lenses (control fitting approach); Device: Test Lenses (test fitting approach)

INTERVENTIONS:
Device: Control Lenses (control fitting approach) — Daily wear multifocal lenses for 1 week
Device: Test Lenses (test fitting approach) — Daily wear multifocal lenses for 1 week

SUMMARY:
The purpose of this study was to compare the clinical performance of two fitting approaches for multifocal contact lenses.

DETAILED DESCRIPTION:
This was a prospective, cross-over, double-masked (participants and investigator), randomized order of testing study. It compared two fitting approaches for silicone hydrogel multifocal contact lenses to assess which method achieved greater vision satisfaction and performance.

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years old;
* Have read and understood the Participant Information Sheet;
* Have read, signed and dated the Informed Consent;
* Best corrected visual acuity of at least 20/25 in each eye;
* Have normal eyes with the exception of the need for visual correction;
* Current multifocal contact lens wearer;
* Spectacle refraction:

Distance: Sphere: -6.00D to + 4.00D Astigmatism: 0.00D to -0.75D Near Addition: Established Presbyopes: +1.50D & +1.75D

* Be willing and able to adhere to the instructions set in the clinical protocol and maintain the appointment schedule.

Exclusion Criteria:

* Ocular anterior segment infection, inflammation, abnormality, or active disease that would contraindicate contact lens wear;
* Use of systemic or ocular medications for which contact lens wear could be contraindicated as determined by the investigator;
* Monocular participants (only one eye with functional vision) or participants fit with only one lens;
* Any moderate or severe ocular condition observed during the slit-lamp examination at the enrolment visit;
* History of herpetic keratitis, ocular surgery or irregular cornea;
* Known pregnancy or lactation during the study period;
* Enrolment of the investigator or his/her staff, family members of the investigator, family members of the investigator's staff, or individuals living in the households of these individuals.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Guillon, PhD, FCOptom, Principal Investigator — Ocular Technology Group - International
Locations (1):
- Ocular Technology Group - International, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-five participants were screened and subsequently enrolled in the study.
Groups:
- Control Lenses, Then Test Lenses: Participants first wore Control Lenses for 1 week (Period 1) and then wore Test Lenses for 1 week (Period 2)
- Test Lenses, Then Control Lenses: Participants first wore Test Lenses for 1 week (Period 1) and then wore Control Lenses for 1 week (Period 2)
Period: Period 1 (One Week)
Arm/Group | Control Lenses, Then Test Lenses | Test Lenses, Then Control Lenses
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: Period 2 (One Week)
Arm/Group | Control Lenses, Then Test Lenses | Test Lenses, Then Control Lenses
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: Includes all study participants.
Arm/Group | Overall Study Population
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall Vision Satisfaction
Description: Overall vision satisfaction for each lens was measured on a 0-100 point Visual Analog Scale (VAS), where 0=Extremely Unsatisfied and 100=Extremely Satisfied
Time Frame: One week
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Lenses: Participants that received Control Lenses during either the first or second period of the study.
- Test Lenses: Participants that received Test Lenses during either the first or second period of the study.
Arm/Group | Control Lenses | Test Lenses
Number analyzed (Participants) | 25 | 25
score on a scale | 78.6 (18.3) | 83.5 (14.9)

2. Primary Outcome: Overall Lens Preference
Description: Participants selected their preferred lens fitting approach from options - 'Control', 'Test', or 'No Preference'
Time Frame: Two weeks
Measure: Count of Participants; unit: Participants
Groups:
- Contact Lens Overall Preference: All participants that completed the study.
Arm/Group | Contact Lens Overall Preference
Number analyzed (Participants) | 25
Participants
  Control Lenses | 10
  Test Lenses | 11
  No Preference | 4

3. Secondary Outcome: Overall Binocular Visual Acuity Index
Description: Mean binocular visual performance for each lens was measured by timed logMAR charts. Overall binocular logMAR visual acuity index was calculated by taking the mean of distance and near visual acuities
Time Frame: One week
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Control Lenses | Test Lenses
Number analyzed (Participants) | 25 | 25
logMAR | 0.12 (0.04) | 0.09 (0.05)

4. Secondary Outcome: Number of Contact Lenses
Description: This measured the ease of fitting each contact lens. It counted the number of contact lenses (pair), selected as per the fitting guide, used to determine the final contact lens to dispense.
Time Frame: One week
Measure: Mean (Standard Error); unit: number of contact lenses (pair)
Arm/Group | Control Lenses | Test Lenses
Number analyzed (Participants) | 25 | 25
number of contact lenses (pair) | 1 (0) | 1 (0)

ADVERSE EVENTS:
Time Frame: Duration of the study, approximately 2 weeks
Arm/Group | Control Lenses | Test Lenses
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/46/NCT05734846/Prot_SAP_000.pdf